CLINICAL TRIAL: NCT05736770
Title: Effect of Pre-operative Respiratory Rehabilitation on Post- Operative Outcomes in Coronary Artery Bypass Graft Patients
Brief Title: Pre-operative Respiratory Rehabilitation in Coronary Artery Bypass Graft Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah/RCRS/REC/ 01378
Record Dates: First submitted 2023-01-13; First posted 2023-02-21 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Respiratory Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory rehabilitation and out of bed mobilization group (Experimental): The Respiratory rehabilitation and out of bed mobilization group will perform 4 exercises.
  Interventions: Other: Respiratory rehabilitation and out of bed mobilization
- Conventional exercise program group (Active Comparator): The conventional exercises program will perform conventional exercises
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: Respiratory rehabilitation and out of bed mobilization — The Respiratory rehabilitation and out of bed mobilization group will perform following exercises: pre operative out of bed mobilization, active cycle breathing techniques, forced expiratory technique and volume based incentive spirometery
  Arms: Respiratory rehabilitation and out of bed mobilization group
Other: conventional treatment — The conventional exercise program group will perform :Flow based Incentive spirometery, Chest percussion if needed
  Arms: Conventional exercise program group

SUMMARY:
To compare the effects of conventional preoperative respiratory rehabilitation and specific preoperative respiratory rehabilitation program on pulmonary functions in coronary artery bypass graft patients.

DETAILED DESCRIPTION:
After cardiac surgeries many postoperative changes occur that lead to pulmonary complication such as respiratory changes, functional capacity of lungs and gaseous changes that leads to hypoxemia and ischemic injury of lungs. CABG, although a successful procedure, post operative pulmonary complications still pursue a big challenge to the health and fitness of the patients. Although post operative complications have been managed in in-patient setup post CABG, there are pre-operative measures on the rise to prevent the complications to occur after CABG.

This study will contribute in describing the rate of improvement in pulmonary functions with rehabilitation program including preoperative out of bed mobilization, active cycle breathing techniques, forced expiratory technique and volume-based incentive spirometry as compared to the conventional treatment of flow-based incentive spirometry and chest percussion in prevention of post operative pulmonary complications occurring after CABG leading to delayed recovery of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective Coronary Artery Bypass Grafting (CABG) surgery for Triple vessel coronary artery disease (TVCAD), double vessel coronary artery disease (DVCAD), single vessel coronary artery disease (SVCAD) and left main stem (LMS) disease.
* Patients who cover at least 400 steps on 6-minute walk test.
* Patients with ejection fraction 45% or more

Exclusion Criteria:

* Acute ailments i.e., patient's cardiac condition deteriorating.
* Cardiac emergency (shock, acute MI)
* Presence of neurological disorders e.g., altered state of consciousness, paralysis.
* Redo surgeries
* Any musculoskeletal disorder e.g., amputation of limb, problems of balance and risks of fall, muscles weakness grade 3 or less, osteoporosis; leading to limitation in exercise.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | 4th postoperative day of coronary artery bypass graft (CABG)
  The Forced Expiratory Volume in 1 Second parameter measures the volume of air that was exhaled into the mouthpiece in the first second after a full inhalation. The normal test values range between 80% and 120% of the average (predicted) values.
Forced Vital Capacity (FVC) | 4th postoperative day of coronary artery bypass graft (CABG)
  Forced Vital Capacity measures the total volume of air that you were able to blow forcefully into the mouthpiece following a full inhalation
Ratio of Forced expiratory volume in 1 second and Forced Vital Capacity (FEV1/FVC) | 4th postoperative day of coronary artery bypass graft (CABG)
  FEV1/FVC: The FEV1/FVC Ratio (FEV1%) parameter is calculated by dividing the measured FEV1 value by the measured FVC value. In healthy adults of the same gender, height, and age, the normal Predicted percentage should be between 70% and 85.

SECONDARY OUTCOMES:
6-minute walk test (6MWT) | 4th postoperative day of coronary artery bypass graft (CABG)
  six minutes walk test (6MWT) is test used to measure functional exercise capacity of patients with cardiovascular and/or pulmonary disease. In this test, patient performs walk for 6 minutes while time being counted on stopwatch. The patient can take rest between the walk, but the timer keeps on running and the rest period is counted. At the end of the test, patient's level of exertion is noted, and the distance measured is recorded. The 6MWT distance values for a healthy person are 400-700m.
Borg scale | 4th postoperative day of coronary artery bypass graft (CABG)
  The Borg Rating of Perceived Exertion (RPE) scale is a tool for measuring an individual's effort and exertion, breathlessness and fatigue during physical work. Patients are asked to tell the whole feeling of exertion including leg pain and shortness of breath and it is marked on a number from 6-20, where 6 indicates "no exertion at all" and 20 indicates "maximal exertion".

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ali Awan, MS-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Muhammad ali awan, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No